CLINICAL TRIAL: NCT04832672
Title: The Optimal Sequence of Intracranial Radiotherapy Compared to Systematic Tyrosine Kinase Inhibitors for Gene-driven Brain Metastases in Targeted Treatment Era
Brief Title: Sequence of Radiation and Targeted Therapy in Brain Metastases
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianping Xiao, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC-005269
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: The Optimal Sequence of Radiotherapy and Systematic Tyrosine Kinase Inhibitors in Treating Brain Metastases
Keywords: Brain metastases; Radiotherapy; Targeted therapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The upfront radiotherapy group
- The upfront targeted-therapy group

SUMMARY:
The investigators conducted a single institutional, retrospective cohort study to demonstrate the appropriate treatment strategy of upfront intracranial radiotherapy or upfront targeted therapy in patients with brain metastases, including an assessment of its feasibility and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Had histologically proven primary cancer.
* Had newly diagnosed brain metastases in contrast-enhanced MRI.
* Brain metastases focus should be measurable.
* All the patients should safely receive radiotherapy and/or systematic tyrosine kinase inhibitors.
* Karnofsky performance score (KPS) ≥60 or KPS ≥40, but only caused by brain metastases.

Exclusion Criteria:

* Patients with prior intracranial local treatments, such as surgery and radiotherapy without dose prescription in detail
* Patients with leptomeningeal metastases at first diagnosis.
* Had synchronous or metachronous malignancies that might affect survival.
* Had severe systemic diseases, abnormal conditions that might lead to incoordinate behavior during the implementation of clinical measures.
* Had incomplete sociodemographic and/or clinicopathologic baseline data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent hypofractionated stereotactic radiotherapy planning at our institution from October 2010 to October 2020
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Intracranial progression-free survival | The interval from the start of initial intracranial treatment to first documented intracranial progression, or date of death from any cause, whichever came first, assessed up to 3 to 5 years
  The survival time of patients before any intracranial progression

SECONDARY OUTCOMES:
Overall survival | The time from the date of initial intracranial treatment until death from any cause or censored on the last follow-up, whichever came first, assessed up to 3 to 5 years
  The survival time of patients
Brain metastasis-specific survival | The interval from the start of initial intracranial treatment to death from brain metastases or censored on the last follow-up, whichever came first, assessed up to 3 to 5 years
  The survival time of patients dead from brain metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yang S, Xiao J, Liu Q, Zhang Y, Bi N, Huang X, Chen X, Wang K, Ma Y, Deng L, Wang W, Zhao R, Li J, Yi J, Wang S, Li Y. The Sequence of Intracranial Radiotherapy and Systemic Treatment With Tyrosine Kinase Inhibitors for Gene-Driven Non-Small Cell Lung Cancer Brain Metastases in the Targeted Treatment Era: A 10-Year Single-Center Experience. Front Oncol. 2021 Oct 14;11:732883. doi: 10.3389/fonc.2021.732883. eCollection 2021. PMID 34722275